CLINICAL TRIAL: NCT00906971
Title: Physiotherapeutic Intervention in Children With Chronic Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Carlos Andre Gomes Silva, Master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: posca-832
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Constipation
Keywords: Physical Therapy; Chronic Functional Constipation; Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laxatives (Active Comparator): Magnesium hydroxide for which the dosage varied according to individual needs (a minimum of 2 ml/kg), and received guidance regarding fiber-rich foods, water and toilet training. Patients attended weekly consultations with a pediatric gastroenterologist.
  Interventions: Other: diaphragmatic breathing, isometric training of the abdominal muscles and abdominal massage

INTERVENTIONS:
Other: diaphragmatic breathing, isometric training of the abdominal muscles and abdominal massage — Exercises will be conducted by one physiotherapist. A one-minute rest period will be observed between each series. Isometric training of the abdominal muscles: This will consist of a contraction of the upper abdomen muscle and diaphragm and the simultaneous relaxation of the lower abdomen. Training will be carried out in two manners: with the patient lying in a left lateral decubitus position with the hip and knee flexed at 90º and sitting. Breathing exercises: With the patient in a seated position, with one hand placed on the abdomen and the other on the thorax, and will be instructed to breath in slowly,. Two series will be completed, with ten repetitions. Abdominal massage: The physiotherapist will perform slow circular clockwise movements, along the line of the colon, with a regular tennis ball, remaining on each point for one minute, beginning with the ascending colon moving in the direction of the sigmoid colon.

SUMMARY:
The purpose of this study is to determine whether physiotherapy is effective in the treatment of the chronic functional constipation in children.

DETAILED DESCRIPTION:
1) INTRODUCTION

Chronic functional constipation (CFC) is a common problem in the pediatric population, affecting approximately 25% of those seeking specialized medical care. The complaint is multifactorial, involving environmental, psychological and physiological factors, which interact with the brain-gut axis, but the retention of stools secondary to the pain-restraint cycle, associated to the fear and anxiety of the resulting bowel movement, is important in the development and management of CFC.

Difficulties involved in the management of CFC are common. Conventional treatment includes educational measures, disimpaction, laxatives and an increased fiber intake. However, these measures have not necessarily been beneficial for all cases, with a cure ratio of between 50 and 60%, and around one third of all patients become long-term sufferers of constipation.

The muscles of the intestine contribute to atonic constipation - sluggish or flaccid muscles in the bowel or rectum, or spasticity - increased muscle tone due to emotional stress. These two factors are both present in patients with CFC. Bowel movement depends on the interlinked functions of abdominal muscles, the pelvic floor and diaphragmatic breathing: contraction of the diaphragm, abdominal distention resulting from the voluntary relaxation of the abdominal wall and the pelvic floor lead to increased intra-abdominal and peristaltic pressure and relaxation of the external anal sphincter (EAS), thus culminating in bowel movement. Added to which, activity of the parasympathetic autonomic nervous system causes an increase in gastrointestinal motility and relaxation of the sphincters. The superficial and deep abdominal muscles, in addition to the diaphragm and muscles of the pelvic floor, form a single muscle unit that assists regular bowel movement, and should all be worked together in order to stimulate peristalsis. Therefore, a combination of exercises that stimulate and relax the abdominal muscles, indirectly acting on the pelvic floor, coordinated with diaphragmatic breathing, may trigger contraction of the intestinal and rectal muscles, therefore bringing relief to patients with CFC.

Multidisciplinary treatment can complement the conventional treatment of CFC. Physiotherapy exercises for the abdominal muscles and diaphragm plus abdominal massage may reverse any changes brought on by CFC. Retraining the intestinal functions is brought about due to two main effects:

1. mechanical - stimulating colonic movements, improving coordination of the muscles involved in bowel movement, thus encouraging fecal propulsion and increasing abdominal muscle tone;
2. neurological - parasympathetic stimulation increases muscle motility, while sympathetic stimulation reduces anxiety, promoting relaxation and increasing endogenous serotonin, thus reducing discomfort and increasing a sense of well-being. However, little evidence of physiotherapy exercises applied to patients with CFC is available in the literature, and randomized, controlled clinical trials are needed.

The aim of the present study is to assess the effect of muscular training, abdominal massage and diaphragmatic breathing in patients with CFC. The hypothesis is that exercises for training abdominal muscles, a diaphragmatic breathing pattern and abdominal massage increase the frequency of bowel movements and reduce episodes of fecal incontinence in patients with CFC.

2) METHODS

Design overview

A randomized, controlled trial was conducted with two parallel groups. In the physiotherapy group, physiotherapy exercises will be employed (isometric training of the abdominal muscles, diaphragmatic breathing exercises and abdominal massage) together with conventional treatment (disimpaction, when necessary, a high-fiber diet, laxatives and toilet training). Patients in the medication group will be only submitted to conventional treatment. Disimpaction will be conducted with phosphate saline solution (once a day, from one to five days, according to patient needs). During toilet training, the patient will be instructed to sit on the toilet for at least five minutes, with support for the feet, after the three main meals of the day.

Setting and participants

The trial will carried out in the Pediatric Unit at Hospital das Clínicas at Federal University of Pernambuco (UFPE), which provides patients with tertiary health care. Children and adolescents aged between 4 and 18 years take part in the study.

For inclusion in the study, patients will be considered with CFC presented two or more of the following parameters in the basal period, at least once a week, during the previous two-month period, according to Rome III criteria: two or less bowel movements per week, at least one episode of fecal incontinence per week, reports of retentive behavior, episodes of hard stools or pain during bowel movements, presence of a large quantity of stool in the rectum and large diameter stools, which could obstruct the toilet. Exclusion criteria will be patients who take medication that caused constipation, patients with organic causes and children with cognitive problems to perform the protocol. Children aged four to six years were assessed for their ability to complete the physiotherapy exercises. This assessment will consist of a few repetitions of the protocol conducted shorter after completing the forms, where difficulty in completing protocol exercises will considered non-inclusion criteria, so as not to interfere with the results.

Parents or guardians will sign the terms of informed consent after receiving information on the aims and procedures of the study. A specially structured form will apply regarding signs and symptoms of CFC. The study was approved by the Ethics Committee for Research involving human beings at the Centro Integrado de Saúde Amaury de Medeiros (Registration 085/08).

Randomization and interventions

A table of random numbers will be created in the computer by someone not involved in the study, from which will determined the random distribution sequence of the patients. This information will remain the exclusive knowledge of one research assistant, who will use these numbers to allocate patients by order of study entry, immediately after giving their consent to take part. This will only made known to the researchers after statistical analysis.

* Physiotherapy + medication group (Intervention) Physiotherapy exercises will be conducted by one single generalist physiotherapist, specially trained to perform the exercises during the three months prior to the study. Twelve individual sessions will be held twice a week, each lasting forty minutes, and adherence will be confirmed only if patients attended all twelve sessions. A one-minute rest period will be observed between each series of exercises.

  * Isometric training of the abdominal muscles The aim of the training will be to increase intra-abdominal pressure (which compresses the intestines) and the colonic propulsive force during voluntary effort. Considering that there is indirect synergic activation between the pelvic floor muscle and the lower abdominal muscle, the operation of the voluntary isometric contraction of the upper abdomen and the simultaneous relaxation of the lower abdomen improves muscle coordination, relaxation of the pelvic floor and relaxation of the external anal sphincter, thus optimizing bowel movement. This consist of a contraction of the upper abdomen muscle and diaphragm and the simultaneous relaxation of the lower abdomen, under the supervision of the physiotherapist. Training will be carried out in two manners: with the patient lying in a left lateral decubitus position with the hip and knee flexed at 90º and sitting. In the lying method, training began with two series of eight contractions and relaxations, into the third week, and then will increase to two series of twelve contractions and relaxations, and will remain so until the sixth week. In the sitting method, training will begin with one series of three contractions and relaxations lasting ten seconds, increasing to five repetitions in the third week, and remaining so until the sixth week. The exercise will considered successfully carried out when a protrusion of the lower abdomen was visible, indicating the simultaneous relaxation of the lower abdomen and the pelvic floor, from which point the series was initiated.
  * Breathing exercises The aim was to achieve a regular pattern of abdominal breathing and strengthen the abdominal muscle, improving coordination between breathing, the abdominal and anal muscles and colonic propulsion. Standard diaphragmatic breathing will achieve with a modified exercise, under the supervision of the physiotherapist, with the patient in a seated position, with one hand placed on the abdomen and the other on the thorax, and will be instructed to breath in slowly, deeply and progressively for 6 to 8 seconds, retain the air for 10 seconds and exhale slowly for 6 to 8 seconds. Two series will be completed, with ten repetitions, and the exercise was considered successfully performed when greater mobility of the hand placed on the abdomen achieves, compared to minimal or no mobility of the hand on the thorax, from which point the series was initiated.
  * Abdominal massage The aim will be perform propulsive abdominal massage to promote colonic and rectal motility, and train the intestinal function and bowel movement. The physiotherapist will perform slow circular clockwise movements, along the line of the colon, applying constant moderate pressure to the abdomen with a regular tennis ball, remaining on each point for one minute, beginning with the ascending colon moving in the direction of the sigmoid colon.
  * Medication and guidance Patients will use a laxative (magnesium hydroxide), for which the dosage will vary according to individual needs (a minimum of 2 ml/kg), and will receive guidance regarding fiber-rich foods, water and toilet training. Patients will attend weekly consultations with a pediatric gastroenterologist, who will be unaware of which patients belonged to which treatment group, since patients were only receiving clinical follow-up.
* Medication Group (Control) Patients in this group will be monitored on a weekly basis by a pediatric gastroenterologist, who will be unaware of which patients belonged to which treatment group, since patients were only receiving clinical follow-up. All patients will be prescribed a laxative (magnesium hydroxide), for which the dosage varied according to individual needs (a minimum of 2 ml/kg), and will receive guidance regarding fiber-rich foods, water and toilet training, under the same conditions as patients in the intervention group.

Sample size Since there are no other similar studies, the sample was calculated from a study that instructed children to achieve bowel movements sitting on the toilet. A reduction was encountered of 80% in fecal incontinence in the intervention group and 55% in the control group. The effect on the reduction of fecal incontinence (< one/week) was estimated at 25% in favor of the intervention. Epi-Info 6.04 was employed, using p=5% power=80%, which resulted in 72 participants.

Outcomes and follow-up The frequency of bowel movement and retentive fecal incontinence will be the primary outcome measures. Pain and increased effort for bowel movement, consistency of stools and retentive behavior will be secondary outcome measures.

During follow-up, parents or guardians will keep a diary describing the intestinal habits of the children. These data will be checked and handed in weekly to the research assistant.

Statistical analysis Statistical analysis to compare the two groups at the end of the follow-up period with regard to the primary and secondary outcome measures will be blind, by intention-to-treat, considering loss of follow-up as treatment failure. In such cases, at the end of the follow-up period, the frequency of bowel movement and fecal incontinence will be recorded, as well as the response to other variables, reported at the beginning of the study. The chi-squared test will be used for proportions and the Student t-test for numerical variations with normal distribution (the Bartlett test was used to verify the homogeneity of the variance). The Mann-Whitney test will be used for numerical variables with non-normal distribution. Statistical significance will set at p<0,05. All analysis will be performed using the Epi-Info™, version 6.04d (CDC - Center of Disease Control and Prevention, Atlanta, USA and WHO World Health Organization, Geneva, swirtzerland).

An intragroup treatment additional exploratory analysis will be also conducted to assess the function of retentive behaviour and fear of bowel movement in the frequency of bowel movement at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Less than 2 per week defecation
* Fecal incontinence
* Retentive behavior
* Pain at defecation and
* Hard stools

Exclusion Criteria:

* Medication use (calcium, antacid, diuretic and hematinic)
* Organic causes (spina bifid, hypothyroidism, hirschusprung disease, developmental delay neuropsychomotor, kidney disease and metabolic diseases)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital's Clinical - UFPE, Recife, Pernambuco, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was carried out in the Pediatric Unit at Hospital das Clínicas at Federal University of Pernambuco (UFPE) between May 2009 and May 2012.
Groups:
- Medication: Magnesium hydroxide for which the dosage varied according to individual needs (a minimum of 2 ml/kg), and received guidance regarding fiber-rich foods, water and toilet training. Patients attended weekly consultations with a pediatric gastroenterologist.
- Physiotherapy + Medication: Physiotherapy exercises were conducted by one single generalist physiotherapist, specially trained to perform the exercises during the three months prior to the study. Twelve individual sessions were held twice a week, each lasting forty minutes, and adherence was confirmed only if patients attended all twelve sessions. A one-minute rest period was observed between each series of exercises.
Period: Overall Study
Arm/Group | Medication | Physiotherapy + Medication
Started | 36 | 36
Completed | 28 | 33
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication | Physiotherapy + Medication | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Customized [Number; unit: participants]
  4 >= 10 years | 20 | 25 | 45
  11 >= 18 years | 16 | 11 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 14 | 16 | 30
Frequency of defecations [Mean (Standard Deviation); unit: days/week] | 2.9 (2.0) | 2.9 (2.3) | 2.9 (2.2)
Retentive fecal incontinence [Mean (Standard Deviation); unit: days/week] | 3.5 (2.6) | 3.6 (2.8) | 3.5 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Defecation.
Description: The patients (or their parents) received a bowel diary and they fulfilled about frequency of defecation weekly.
Time Frame: six weeks
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Medication | Physiotherapy + Medication
Number analyzed (Participants) | 36 | 36
days/week | 3.9 (2.0) | 5.1 (2.1)
Statistical Analysis 1: Comparison: Medication vs Physiotherapy + Medication; Test type: Non-Inferiority or Equivalence — Statistical analysis to compare the two groups at the end of the follow-up period with regard to the primary outcome measures was blind, by intention-to-treat, considering loss of follow-up as treatment failure. In such cases, at the end of the follow-up period, the frequency of defecations was recorded; p < 0.05, t-test, 1 sided; The Mann-Whitney test was used for numerical variables with non-normal distribution

2. Primary Outcome: Retentive Fecal Incontinence.
Description: Retentive fecal incontinence is the lose of fecal while the patient tries to avoid the bowel movement.
  The patients (or their parents) received a bowel diary and they fulfilled about frequency of episodes of retentive fecal incontinence weekly.
Time Frame: six weeks
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Medication | Physiotherapy + Medication
Number analyzed (Participants) | 36 | 36
days/week | 3.0 (2.1) | 3.6 (1.9)
Statistical Analysis 1: Comparison: Medication vs Physiotherapy + Medication; Test type: Non-Inferiority or Equivalence — Statistical analysis to compare the two groups at the end of the follow-up period with regard to the primary outcome measures was blind, by intention-to-treat, considering loss of follow-up as treatment failure. In such cases, at the end of the follow-up period, the frequency of fecal incontinence was recorded reported at the beginning of the study; p > 0.05, t-test, 1 sided; The Mann-Whitney test was used for numerical variables with non-normal distribution

ADVERSE EVENTS:
Arm/Group | Medication | Physiotherapy + Medication
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

LIMITATIONS AND CAVEATS:
The study was not designed to assess if a longer period of physiotherapy using these exercises could bring more clinical benefits to bowel habits, therefore, further studies should be undertaken to assess longer treatment periods, of 6 to 12 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No